CLINICAL TRIAL: NCT00116545
Title: TART - Troglitazone Atherosclerosis Regression Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Parke-Davis (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG0028; 991-081-00
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2005-06

CONDITIONS: Atherosclerosis; Diabetes Mellitus
Keywords: IDDM; Insulin; cardiovascular disease
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus; Diabetes Mellitus, Type 1; Insulin Resistance; Cardiovascular Diseases | interventions — Troglitazone

INTERVENTIONS:
Drug: troglitazone

SUMMARY:
The purpose of this study is to determine if troglitazone reduces the progression of early preintrusive carotid atherosclerosis in insulin-requiring diabetes patients.

DETAILED DESCRIPTION:
Insulin resistance and hyperinsulinism appear to be important risk factors for the development of atherosclerosis in diabetes patients. The atherogenic potential of insulin has been shown to improve cholesterol and may have an effect on the thickness and structure of the arterial wall. Troglitazone is an oral diabetic agent that treats insulin resistance. Based on the initial data available, it would appear that troglitazone may be effective in both glycemic control and improved atherosclerosis risk in diabetes patients. This study will compare the effects of troglitazone to placebo in insulin-requiring diabetes patients on both glycemic control and progression of atherosclerosis.

A total of 288 men and women 30 to 70 years of age with insulin-treated diabetes were recruited and entered an 8 week run-in phase to stabilize diet, exercise, insulin dose and glucose levels. Upon successful completion of the run-in phase, all patients were randomized into one of two groups to receive either troglitazone 400mg/day or a matching placebo while continuing with diet and exercise regimens and insulin dose to maintain pre-meal glucose levels between 100 to 150 mg/dL.

Follow up visits occurred every 2 weeks for 2 months, every 4 weeks for 2 months, then every 8 weeks for the remainder of the 2-year trial. The progression of atherosclerosis was measured by ultrasonography at baseline and every 6 months throughout the 2 years of randomized treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 30-70 years
* Diabetes: fasting glucose over 140 mg/dL but under 350 mg/dL on at least 2 occasions
* At least 30 years of age at onset of diabetes
* Metabolic control and management requiring insulin without other anti-diabetic medications
* Willingness to sign informed consent

Exclusion Criteria:

* Known sensitivity to troglitazone or other thiazolidinediones
* For premenopausal females: pregnancy, breastfeeding, unwilling to use effective contraception for the duration of the trial
* Active liver disease or hepatic dysfunction; renal dysfunction; high blood pressure; major vascular events within 6 months prior to randomization; untreated hypothyroidism or uncured hyperthyroidism; other severe or unstable disease within 5 years of randomization
* Medical illness that may require oral or parenteral glucocorticoid therapy
* Physical disability that would interfere with diabetes self-management
* Untreated or unstable diabetic retinopathy
* History of insulin allergy
* Present or recent history of alcohol intake over 5 drinks per day or substance abuse
* Participation in another clinical trial
* Currently taking nicotinic acid

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288
Dates: Start 1997-01; Primary Completion 2000-04 (Actual); Study Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
rate of change of the right distal common carotid artery far wall intima-media thickness (IMT) measured every 6 months
flow mediated brachial artery vasoactivity

SECONDARY OUTCOMES:
carbohydrate and lipid metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Howard N. Hodis, MD, Principal Investigator — University of Southern California, Atherosclerosis Research Unit, Division of Cardiovascular Medicine, Department of Medicine
Locations (1):
- Atherosclerosis Research Unit, Division of Cardiovascular Medicine, Department of Medicine, Los Angeles, California, United States